CLINICAL TRIAL: NCT05226377
Title: High Atherogenic Index of Plasma At-admission of COVID-19 Patients Can Predict Upcoming Cardiac Morbidity and Mortality in Non-Cardiac Patients
Brief Title: Relation Between Atherogenic Index of COVID-19 and Upcoming Cardiac Morbidity and Mortality in Non-Cardiac Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Fayez Al-kassas, lecturer of Cardiology, Tanta University
Other Study IDs: 35069/11/21
Record Dates: First submitted 2022-01-21; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Atherogenic Index of Plasma — - The atherogenic index of plasma (AIP) is defined as the base 10 logarithms of the ratio of plasma triglyceride (TG) to high-density lipoprotein cholesterol (HDL-c) (17). AIP was employed as a predictor of cardiac risk (CR) with values of -0.3 to 0.1 are associated with low, values of 0.1-0.24 are associated with the medium, and values above 0.24 with high CR

SUMMARY:
Plasma lipids levels were estimated and the Atherogenic Index of Plasma (AIP) was computed in 302 COVID confirmed patients. Patients were evaluated using the COVID-GRAM (CG) critical illness score and during a hospital stay the rates of admission to intensive care unit (ICU), development of cardiac insults, and need for admission to cardiac ICU (CCU) and its outcome were determined.

DETAILED DESCRIPTION:
All patients were admitted to the quarantine department at Tanta University hospital and quarantine hospitals at Al-Gharbia governorate with a diagnosis of SERS-CoV-19 infection that was confirmed by having positive nasopharyngeal swab for SARS-CoV-2 using reverse transcriptase-polymerase chain reaction (RT-PCR). The study protocol was approved by the Local Ethical Committee according to instructions of the Ministry of Health and written informed consents were signed by all enrolled patients or their nearest relative.

Using the strict personal protective equipment, patients were clinically examined for collection of the demographic data age, sex, weight and height, history taking especially past and/or present history of diabetes mellitus (DM), hypertension, cardiac diseases, hypercoagulability events, chest, liver or kidney diseases or endocrinopathy. BMI was calculated in kg/m2 as weight (kg)/height (m2) (14) and was graded according to the guidelines of WHO (15). The chest was examined clinically and CT imaging was performed to assess the disease severity.

Clinical parameters

1. COVID-19 disease severity grading
2. COVID-GRAM Critical Illness Risk Score
3. Atherogenic index of plasma (AIP)

Laboratory investigations A- Routine lab investigations included estimation of random blood glucose, complete blood count and serum levels of urea, creatinine, liver enzymes, and total and direct bilirubin B- Investigations for evaluation of SARS-CoV-2 infection severity including estimation of serum C-reactive protein, interleukin-6, lactate dehydrogenase, D-dimer levels.

C- Estimation of a plasma lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Only non-cardiac patients with confirmed COVID-19 disease who had mild-to-severe COVID disease according to the guidelines of the National Institutes of Health admitted to quarantine hospitals and free of exclusion criteria were enrolled in the study. Patients were categorized according to disease severity into mild, moderate, and severe.

Exclusion Criteria:

* Patients presented by COVID disease of critical severity that necessitated admission to ICU at time of hospital attendance, admission to ICU for any other indication, presence of a history of cardiac diseases, previous cardiothoracic or chest surgery for any indication, BMI of ≥35 kg/m2, presence of endocrinopathy, preexisting autoimmune diseases, current maintenance on immunosuppressive drugs, malignancy elsewhere in body organs, refusal to sign the written consent to receive the study protocol or death just on admission or before completion of the diagnostic protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: COVID confirmed patients free of Cardiac Diseases evaluated Clinically by laboratory investigations
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | two weeks
  Development of new cardiac insult
Mortality | two weeks
  Death of patients due to new cardiac insult

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt